CLINICAL TRIAL: NCT04467385
Title: Effects Of Virtual Reality Training With Sensory Integration On The Gross Motor Functions Of Lower Limb In Spastic Diplegic Cerebral Palsy.
Brief Title: Virtual Reality Training With Sensory Integration On The Gross Motor Functions Of Lower Limb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00557 Sannia Batool
Record Dates: First submitted 2020-03-18; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Cerebral Palsy Spastic Diplegia
Keywords: Virtual Reality; Spastic Diplegic Cerebral Palsy; Sensory Integration
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Virtual Reality training(VR) + Sensory Integration therapy + conventional therapy
  Interventions: Other: VR training + Sensory Integration therapy + conventional therapy
- Control Group (Experimental): VR training + conventional therapy
  Interventions: Other: VR training + conventional therapy

INTERVENTIONS:
Other: VR training + Sensory Integration therapy + conventional therapy — After the baseline assessment,
  * Coconut ShootersVR - 5 min/day
  * Ninja flipVR - 5 min/day.
  * Sensory integration training include Exercises on BOSU ball and mini-trampoline. It will involve:
  * Passive bouncing with child standing with his/her feet shoulder width apart for 2.5 and 2.5 minutes on both.
  * Active bouncing (the child bounces and therapist will control the rate) for 2.5 and 2.5 minutes on both.
  * Mini-squat exercises with feet apart and feet together for 2.5 and 2.5 minutes on both.
  * Conventional exercises include:
    * passive stretching exercises for the hip flexors, hip adductors, hamstring, and calf muscle; stretching will be applied for 30 sec with 30 sec rest for each muscle group within pain limit.
    * Strengthening of abdominal and back muscles, hip abductions and knee joint extensors and ankle dorsiflexors will be performed.
  Arms: Experimental Group
Other: VR training + conventional therapy — After the baseline assessment,
  * The Your Shape: Fitness Evolved 2012TM game is selected for VR training (walking and walking with obstacles) for 8 min
  * Coconut ShootersVR - 8 min/day
  * Ninja flipVR - 8 min/day
  * Conventional Therapy - 20 min per day
    * Passive stretching exercises for the hip flexors, hip adductors, hamstring, and calf muscle; stretching will be applied for 30 sec with 30 sec rest 3-5 times for each muscle group within pain limit.
    * Strengthening of abdominal and back muscles, hip abductions and knee joint extensors and ankle dorsiflexors will be performed.
  Arms: Control Group

SUMMARY:
The objectives of this study are To determine the effect of virtual reality on balance and gross motor functions of the lower limb in spastic diplegic cerebral palsy. To determine the effect of virtual reality with sensory input on balance and gross motor functions of the lower limb in spastic diplegic cerebral palsy. To compare the effects of virtual reality training with and without sensory input on balance and gross motor functions of the lower limb in spastic diplegic CP. Its is a Randomized control trial (RCT) done at Physiotherapy department of Railway General Hospital Rawalpindi and National Institute of rehabilitation Medicine.44 individuals (calculated using epi tool) 22 individuals in each group. Individuals who met the inclusion criteria will be included in this study. All participants will go through randomization and divided into two groups Experimental and Control groups. Pre-intervention assessment is made for both groups. Then intervention will be applied to both groups. estimated time of treatment protocol will be 40 min/day, 1 time / d, 3 times/week for 6 weeks. Subjects will be evaluated at baseline, then 3rd week and 6th-week assessment will be the final

DETAILED DESCRIPTION:
Cerebral Palsy(CP) is a common non-progressive disorder that occurs due to any injury or aberration to the developing central nervous system. It refers to the disorders that stem from primary brain lesion leading to musculoskeletal and nervous abnormalities in the pediatric population. Cerebral palsy has a global incidence of 1-3.5 cases per 1000 live births. The most prevalent type is spastic diplegia which occurs in 30-40% of spastic cerebral palsy. According to motor impairment, it is classified into spastic, dyskinetic and ataxic cerebral palsy. The children with cerebral palsy have very poor control of voluntary muscle activity. Therefore training of selective motor control in children with cerebral palsy is an important part of physiotherapy intervention. Children are often not amenable to the conventional exercise program but studies have demonstrated that children show high interest and stimulation to virtual reality training. Virtual reality is a virtual environment system that enables a person to witness situations and actions similar to real-life. Therapists use Virtual reality systems to create a fascinating environment to gain targeted therapeutic goals. Sensory integration, on the other hand, is a therapeutic approach that involves active therapy and activities involving graded sensory experiences. It provides keen proprioceptive and tactile experiences. Sensory integration therapy usually involves balls, rolls, hammock, trampolines and altering surfaces. Children with spastic diplegia have gross and fine motor, sensory, cognitive impairments. This results in reduced ability to adjust the body and balance it with movements. Postural control demands active sensorimotor control. Exercise with mini-trampoline is designed for balance training to improve static and dynamic balance and postural adjustment in children with spastic diplegia. According to a study in 2016, Virtual reality training can effectively improve the gross motor function of the lower limbs in children with spastic diplegia in comparison to conventional therapy. As claimed by a study in, 2006 VR training in combination with conventional exercise therapy in spastic CP improves exercise compliance and enhance exercise effectiveness. It is a simple and executable approach which can be used by any skilled therapist as an independent treatment method to improve the outcome.

According to a study, sensory integration therapy had a measurable effect in children with spastic diplegic cerebral palsy who suffer from a sensory-motor deficit. A study observed the effects of sensory integration therapy in children with cerebral palsy and concluded that sensory integration therapy has a positive effect on gross motor function in spastic diplegic CP in sitting and standing positions. Whereas, the control group with only home exercise program showed no significant improvement.In 2018 compared the effects of rebound exercises and simple balance training on balance of spastic diplegic children. The assessments suggested that balance was improved in both groups but the group under study showed a significant difference and concluded that rebound exercises improve the balance and postural control. The past research records are evident that therapists have worked with either Virtual reality training or Sensory integration therapy for the rehabilitation of Spastic Diplegic children. The two protocols have not been complimented for rehabilitation. So the aim of this study is to observe and determine the combined effect of these two treatment protocols to get the results and improve the gross motor function in lower limbs of CP children.

ELIGIBILITY:
Inclusion Criteria:

* Diplegic CP children aged 5-12 years
* Gross motor function classification system System (GMFCS) I - II
* Children can be independent Walking distance >5 meters
* Spasticity of lower limb < 3 ..
* A child able to understand command and can play VR games.

Exclusion Criteria:

* Any Bone and joint diseases
* Epilepsy
* Mental illness
* Mental retardation etc. cannot be matched with the completion of the experiment.
* Any history of taking anticonvulsant drugs or muscle relaxants.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Pediatric Balance Scale (PBS): | Changes from baseline to 6th month
  Pediatric Balance Scale (PBS) is a modification of Berg Balance Scale was developed as a balance measure for children with mild to moderate motor impairments.
Gross Motor Function Measure (GMFM-88) | Changes from baseline to 6th month
  Its an 88-item tool for assessing and measuring changes in gross motor function in children with cerebral palsy. It's a four pint scale from 0-3 that indicates the grading of a specified task and the tool is further divided into five categories.
2 min walk Test (2MWT) | Changes from baseline to 6th month
  The Two/2 Minute Walk Test (2 MWT) is a measure of self-paced walking ability and functional capacity. The 2 MWT is a simple measure of the distance a person can walk in two minutes. Rest breaks are allowed if needed. The person is encouraged to walk as fast as they can, safely, for two minutes. Walking aids can be used as needed.

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bumin G, Kayihan H. Effectiveness of two different sensory-integration programmes for children with spastic diplegic cerebral palsy. Disabil Rehabil. 2001 Jun 15;23(9):394-9. doi: 10.1080/09638280010008843. PMID 11394590
- [Background] Lazzari RD, Politti F, Santos CA, Dumont AJ, Rezende FL, Grecco LA, Braun Ferreira LA, Oliveira CS. Effect of a single session of transcranial direct-current stimulation combined with virtual reality training on the balance of children with cerebral palsy: a randomized, controlled, double-blind trial. J Phys Ther Sci. 2015 Mar;27(3):763-8. doi: 10.1589/jpts.27.763. Epub 2015 Mar 31. PMID 25931726
- [Background] Bulekbayeva S, Daribayev Z, Ospanova S, Vento S. Cerebral palsy: a multidisciplinary, integrated approach is essential. Lancet Glob Health. 2017 Apr;5(4):e401. doi: 10.1016/S2214-109X(17)30082-7. No abstract available. PMID 28288745
- [Background] Bryanton C, Bosse J, Brien M, McLean J, McCormick A, Sveistrup H. Feasibility, motivation, and selective motor control: virtual reality compared to conventional home exercise in children with cerebral palsy. Cyberpsychol Behav. 2006 Apr;9(2):123-8. doi: 10.1089/cpb.2006.9.123. PMID 16640463
- [Background] Snider L, Majnemer A, Darsaklis V. Virtual reality as a therapeutic modality for children with cerebral palsy. Dev Neurorehabil. 2010;13(2):120-8. doi: 10.3109/17518420903357753. PMID 20222773
- [Background] Galli M, Cimolin V, Pau M, Leban B, Brunner R, Albertini G. Foot pressure distribution in children with cerebral palsy while standing. Res Dev Disabil. 2015 Jun-Jul;41-42:52-7. doi: 10.1016/j.ridd.2015.05.006. Epub 2015 Jun 6. PMID 26057837
- [Background] Ren K, Gong XM, Zhang R, Chen XH. [Effects of virtual reality training on limb movement in children with spastic diplegia cerebral palsy]. Zhongguo Dang Dai Er Ke Za Zhi. 2016 Oct;18(10):975-979. doi: 10.7499/j.issn.1008-8830.2016.10.011. Chinese. PMID 27751214